CLINICAL TRIAL: NCT03627156
Title: The Effect of Guided Counseling in Improving Dietary Practice, Nutritional Status and Birth Weight of Pregnant Women in West Gojjam Zone, Amhara Region, Ethiopia: A Cluster Randomized Controlled Community Trial
Brief Title: The Effect of Guided Counseling in Improving Dietary Practice, Nutritional Status and Birth Weight of Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahir Dar University (Other)
Responsible Party: Principal Investigator, Yeshalem Mulugeta Demilew, Assistant professor, Bahir Dar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 092/18-04
Record Dates: First submitted 2018-07-12; First posted 2018-08-13 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Counseling
Keywords: Guided counseling; nutrition outcome; Ethiopia; Community trial

STUDY DESIGN:
Intervention Model Description: A two-arm parallel cluster randomized community trial
Who Masked: Outcomes Assessor
Masking Description: outcome assessors are not informed about the intervention and the group to which the intervention is assigned to avoid social desirability bias
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention Arm is an arm to which community-based guided counseling using Health Belief Model and Theory of Planned Behavior will be given.
  Interventions: Behavioral: guided counseling
- Control (No Intervention): Control Arm is an arm to which the intervention will not be implemented.

INTERVENTIONS:
Behavioral: guided counseling — Community-based guided counseling using Health Belief Model and Theory of Planned Behavior is the intervention package for this study.
  Arms: Intervention

SUMMARY:
Poor dietary intake affects maternal wellbeing, fetal growth, and development. However, many pregnant women in Ethiopia have poor dietary intake. To improve the dietary intake of pregnant women, nutrition education is often given at the community level during a home visit and at the health institution during antenatal care. Yet, there is no evidence on the effect of nutrition education on dietary intake, nutritional status, and birth weight in the study area. Hence, the objective of this study was to evaluate the effect of guided counseling in improving dietary practice, nutritional status and birth weight of pregnant women.

A two-arm parallel cluster randomized community trial was conducted among pregnant women in West Gojjam Zone, Amhara region, Ethiopia from May 2019 to May 2019. Baseline data on dietary practice and nutritional status of pregnant women were collected from May to August 2018 (13weeks). Endline data were collected from October 2018 to May 2019. Guided counseling using the health belief model and theory of planned behavior was given in the intervention arm (11 clusters) for 10 months.

Pregnant women were selected using a cluster sampling method. A validated interviewer-administered structured questionnaire was used for collecting data on the study subjects both at the baseline and after the intervention. Data were checked, coded and double entered into Epi-Info version 7.2.2 and exported to SPSS version 23 for statistical analysis. The outcome of the study finding could be useful for health and nutrition policymakers and other concerned bodies in decision making and to design effective intervention strategies to improve dietary practices of pregnant women as a result to prevent malnutrition. 19,553 US dollar was needed to conduct the study.

DETAILED DESCRIPTION:
In the developed countries, pregnant women take relatively adequate and diversified food while pregnant women in the developing countries consume inadequate amount and less diversified diet with very low energy, folate, iron, zinc, and vitamin A content. But, Asian and African pregnant women took more cereals with a small amount of animal products, vegetables, and fruits.

Similarly, the dietary practice of Ethiopian pregnant women has long been an issue of public health concern since almost all pregnant women take inadequate amount of poor quality diet. Their energy and nutrient intake was below the recommended average requirement. In the country, food taboos are highly prevalent; nonetheless, there is a variation on the type of food considered as taboo and the possible reason for food taboo within the country.

In spite of increasing nutrient demand with increasing gestational age, from the literature trend of dietary change was different from country to country and within the country. Pregnant women in developed countries improve their dietary practices with increasing gestational age. However, pregnant women in developing countries experienced "eating down".

Women who had inadequate dietary intake during pregnancy were more likely to develop under-nourishment compared with their counterparts. Under-nourishment in turn associated with intrauterine growth retardation (IUGR), low birth weight (LBW) and premature delivery.

Not only inadequate intake but also excessive consumption of energy-dense foods associated with increases the risk of adverse pregnancy outcomes such as preeclampsia, gestational diabetes mellitus, hemorrhage, cesarean-section delivery, infection, birth trauma, macrosomic infant, delay or failure to lactate, postpartum weight retention.

To improve maternal and child nutrition, the Ethiopian government developed food and nutrition policy, strategy, and programs with guidelines to implement nutrition-specific and sensitive interventions vital to alleviate nutrition problems. In the country, nutrition education is often given to pregnant women at the community and health institution. Yet, pregnant women have insufficient knowledge and poor dietary practice.

Counseling is a series of professional guidance which aims to change the knowledge, attitude, and behavior of an individual. Guided counseling is identified as an effective measure to improve maternal knowledge on nutrition which is the determinant factor of woman's adherence to a healthy dietary practice. Appropriate dietary practice, in turn, improves nutritional status and birth weight of pregnant women. From the literature, the health belief model and theory of planned behavior constructs are effective to improve the dietary practice of pregnant women. In this study, guided counseling refers to professional guidance based on the health belief model and the theory of planned behavior to improve dietary practice, nutritional status, and birth weight.

Hence, the aim of this study was to assess the effect of guided counseling in improving dietary practice, nutritional status and birth weight of pregnant women in West Gojjam Zone. Dietary practice means the dietary intake of pregnant women. Trimester based nutrition counseling was implemented(the women were counseled to increase portion size and frequency of meal with increasing gestational age). The study used the health belief model and theory of planned behavior constructs and counseling card to counsel the women. Besides, a leaflet with appropriate pictures was given to the women to use it at home.

Methods: The study was conducted among pregnant women in West Gojjam Zone, Amhara Region, Ethiopia from May 2018 to May 2019. Baseline data on dietary practice and nutritional status of pregnant women were collected from May to August 20/2018 (13weeks). Endline data were collected from October 2018 to May 2019. Therefore, a time frame to the second, third and fourth objective was 8months. The study used mixed methods design; quantitative and qualitative study and cluster randomized controlled community trial. Single population proportion formula was used to estimate the sample size for objective I while G power 3.1.9.2 software was used to determine the sample size for objective II, III and IV. Respondents were selected using a randomized cluster sampling technique.

Community-based guided counseling using the health belief model and theory of planned behavior was the intervention package for this study. The core contents of guided counseling were the following: increasing frequency of meal (consumption of at least one additional meal in the second and at least two additional meals during the third trimester of pregnancy), increasing portion size with gestational age, using iodized salt, taking iron/folic acid supplement, eating diversified food by giving emphasis to iron-rich foods, taking fruits and vegetables, include animal source foods in the diet (at least two servings per day), reducing heavy workload, taking daytime rest, using malaria prevention methods and health service.

Moreover, the consequence of inadequate dietary intake, susceptibility to the consequence of insufficient die, the severity of the consequence of inadequate meal intake were also parts of the core content of guided counseling. Attitude, subjective norms, self-efficacy, perceived control, intention, knowledge and dietary practice of pregnant women were also assessed before each counseling session. Then, counseling was given based on the identified gap.

The intervention began before 16 weeks of gestation. Each pregnant woman attended 4 counseling sessions. Each counseling session lasting in 30-60 minutes depending on the number of participants (monthly). Leaflet with core messages in Amharic with appropriate picture was prepared and delivered to each pregnant woman in the intervention arm to use it in their home. Three nurses who have a Bachelor of Science and two public health professionals were recruited as counselor and supervisor of counseling intervention, respectively. Women in the control arm received traditional nutrition education given by the existing health system.

The outcomes of the intervention were measured during 36-37 weeks of pregnancy. Birth weights were measured within 48hours after delivery. The first, second and third outcomes of this intervention were dietary practice and nutritional status of the pregnant women, and birth weight, respectively. Data safety have been monitored by the Data Safety Monitoring Board (DSMB). Data were collected by interviewer-administered questionnaires adapted from previous literature and modified based on the local context.

Data on the socio-demographic and obstetric characteristics were collected during the baseline using a structured questionnaire. Whereas, data on women's knowledge about maternal diet, household food security status, dietary practice, Health Belief Model and Theory of Planned Behavior constructs, Mid-Upper Arm Circumference, weight, and blood pressure were collected before and after implementation of the intervention.

The dietary practices of pregnant women were assessed by a food frequency questionnaire. The nutritional status of pregnant women was assessed using the Mid-Upper Arm Circumference measurement.

Six female diploma nurses and three public health professionals were recruited as data collector and supervisor, respectively. Additionally, three laboratory technicians were recruited to confirm pregnancy. Women who took four or more meals a day and have high Women Dietary Diversity Score and Food Variety Score above the mean and high Animal Source Food consumption were considered as having appropriate dietary practice.

Data were entered using Epi Info version 7.2.2 software and analyzed by SPSS version 23 software. Descriptive statistics were computed. Bivariate and multivariable logistic regression analysis was done. A p-value < 0.2 was used as a cut-off point to select variables for the final model. P-values < 0.05 was considered statistically significant.

Pre-intervention and post-intervention differences in women's dietary diversity score, food variety score, animal source food consumption, dietary practice and nutritional status between the intervention and control groups will be analyzed by using paired sample t-test for continuous variables and chi-squared test for the categorical variables. Dietary practice, nutritional status, and birth weight being nested within clusters, hence mixed effects binary logistic regression models, mixed effects linear logistic regression models and mixed effects multinomial logistic regression model will be used to measure the difference in effect on the dietary practice, nutritional status and birth weight between the intervention groups taking into account for clusters and report the Intraclass correlation coefficient, respectively. Cluster level variables will be analyzed as a random effect in the models, whereas the first level predictors will be managed as a fixed effect.

Various measures have been taken to maintain the quality of the research starting from designing the tool to data analysis and interpretation of the result. The questionnaires were adapted and pretested. Three days of intensive training was given to the counselors, data collectors, and supervisors using the training manual. An equal number and non-adjacent clusters for intervention and control group were taken from each Woreda to neutralize the effect of variations if any. Close supervision has been done by supervisors and principal investigator during counseling and data collection.

A cross-sectional phenomenological qualitative study using both key informant interviews and focus group discussions have been used to supplement the quantitative data. Qualitative data was collected until saturation of information. Typical case sampling and extreme sampling technique were used to select the study participants for the key informant interviews and homogeneous sampling for focus group discussions. Semi-structured interview and focus group discussion guides were developed to collect qualitative data.

To assure the quality of data the interviews and facilitation of focus group discussions were done by a principal investigator. To assure trustworthiness triangulation was used in data sources, during data collection and research methodologies. Thematic framework analysis technique will be used to analyze data.

The study was approved by the Institutional Review Board of Bahir Dar University. Written permission was obtained in West Gojjam zone and each Woreda administrators. The intervention was registered in Clinical Trials.gov. Written consent was secured from each participant after explaining the purpose of the study, the right of the participants to withdraw from the study at any time during the study period, potential risk and benefits. Confidentiality has been maintained throughout the study. Undernourished women and women with high blood pressure have been referred to the nearby health institution for treatment. Written consent was secured from individuals who give their picture for leaflet preparation. If the intervention is effective, the project will be implemented in the control area.

ELIGIBILITY:
Inclusion Criteria:

* <16weeks of gestation
* living in the Kebele at least for six months
* has planned to give birth in the study area.

Exclusion criteria:

* Diabetes millitus
* Hypertension

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Dietary practice (dietary intake) | 10 month of intervention
  Improve dietary practice after intervention. Taking more than three meals daily plus the highest tercile of women's dietary diversity score from nine food groups plus the highest tercile of animal source food consumption plus food variety score above the mean

SECONDARY OUTCOMES:
nutritional status | 10 months of intervention
  Improve mid-upper arm circumference (cm) of the pregnant women after intervention.
Birth weight | 10 month of intervention
  Increase in birth weight (gram) after intervention
Dietary practice | 10 weeks (baseline)
  Baseline dietary practice of pregnant women before the implementation of intervention. Taking more than three meals daily plus the highest tercile of women's dietary diversity score from nine food groups plus the highest tercile of animal source food consumption plus food variety score above the mean

CONTACTS AND LOCATIONS:
Overall Officials: Getu Alene, Phd, Study Director — Bahir Dar University
Locations (1):
- Bahir Dar University, Bahir Dar, Ethiopia

IPD SHARING:
Plan to Share IPD: No
I have no plan to share data for other researchers.

REFERENCES:
- [Background] Kanadys WM. Maternal underweight and pregnancy outcome: prospective cohort study. Archives of Perinatal Medicine. 2007;13(3):23-6.
- [Background] Changamire FT, Mwiru RS, Msamanga GI, Spiegelman D, Urassa W, Hertzmark E, Fawzi WW, Peterson KE. Macronutrient and sociodemographic determinants of gestational weight gain among HIV-negative women in Tanzania. Food Nutr Bull. 2014 Mar;35(1):43-50. doi: 10.1177/156482651403500106. PMID 24791578
- [Background] Rolfers SR, Pinna K, Whitney E. Understanding Normal and Clinical Nutrition,eighth edition. Wadsworth: Yolanda Cossio; 2009.
- [Background] WHO Recommendations on Antenatal Care for a Positive Pregnancy Experience. Geneva: World Health Organization; 2016. Available from http://www.ncbi.nlm.nih.gov/books/NBK409108/ PMID 28079998
- [Background] Santiago SE, Park GH, Huffman KJ. Consumption habits of pregnant women and implications for developmental biology: a survey of predominantly Hispanic women in California. Nutr J. 2013 Jul 1;12:91. doi: 10.1186/1475-2891-12-91. PMID 23815874
- [Background] Smedley J, Jancey JM, Dhaliwal S, Zhao Y, Monteiro SM, Howat P. Women's reported health behaviours before and during pregnancy: A retrospective study. Health Education Journal. 2014;73(1):28-40.
- [Background] Lee SE, Talegawkar SA, Merialdi M, Caulfield LE. Dietary intakes of women during pregnancy in low- and middle-income countries. Public Health Nutr. 2013 Aug;16(8):1340-53. doi: 10.1017/S1368980012004417. Epub 2012 Oct 9. PMID 23046556
- [Background] Sun E, Sameera T, Mario M, Laura E. Whate are African Women Eating During Pregnancy? . FASEB Journal. 2011;25:592.
- [Background] Asayehu TT, Lachat C, Henauw S, Gebreyesus SH. Dietary behaviour, food and nutrient intake of women do not change during pregnancy in Southern Ethiopia. Matern Child Nutr. 2017 Apr;13(2):e12343. doi: 10.1111/mcn.12343. Epub 2016 Jul 3. PMID 27373896
- [Background] Fall C. Maternal nutrition: effects on health in the next generation. Indian J Med Res. 2009 Nov;130(5):593-9. PMID 20090113
- [Background] Abu-Saad K, Fraser D. Maternal nutrition and birth outcomes. Epidemiol Rev. 2010;32:5-25. doi: 10.1093/epirev/mxq001. Epub 2010 Mar 17. PMID 20237078
- [Background] Sukhwinder K. Outcomes of prenatal nutrition counseling In developing countries, A Literature Review. 2010
- [Background] Glanz K, Rimer BK, Viswanath K, editors. Health behavior and health education : theory, research, and practice / . 4th ed. San Francisco: Jossey-Bass; 2008.
- [Background] Verbeke W. Impact of communication on consumers' food choices. Proc Nutr Soc. 2008 Aug;67(3):281-8. doi: 10.1017/S0029665108007179. Epub 2008 May 23. PMID 18498672
- [Derived] Demilew YM, Alene GD, Belachew T. Effects of guided counseling during pregnancy on birth weight of newborns in West Gojjam Zone, Ethiopia: a cluster-randomized controlled trial. BMC Pediatr. 2020 Oct 6;20(1):466. doi: 10.1186/s12887-020-02363-8. PMID 33023521
- [Derived] Demilew YM, Alene GD, Belachew T. Effect of guided counseling on dietary practices of pregnant women in West Gojjam Zone, Ethiopia. PLoS One. 2020 May 26;15(5):e0233429. doi: 10.1371/journal.pone.0233429. eCollection 2020. PMID 32453774
- [Derived] Demilew YM, Alene GD, Belachew T. Effect of guided counseling on nutritional status of pregnant women in West Gojjam zone, Ethiopia: a cluster-randomized controlled trial. Nutr J. 2020 Apr 28;19(1):38. doi: 10.1186/s12937-020-00536-w. PMID 32345286